CLINICAL TRIAL: NCT05562570
Title: Exercise Intervention Coupled With Standard Post-cancer Directed Treatment Care to Reduce Chronic Pain in Adolescents and Young Adult Cancer Survivors Who Have Completed Cancer-directed Therapy Less Than One Year
Brief Title: Exercise and Pain in AYACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Smita Dandekar, Principal Investigator, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00020904
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: AYA Cancer Survivors

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity intervention coupled with standard post-cancer directed treatment care group (Experimental)
  Interventions: Behavioral: Physical activity intervention coupled with standard post-cancer directed treatment care
- Standard post-cancer directed treatment care control group (Other)
  Interventions: Other: Standard post-cancer directed treatment care control

INTERVENTIONS:
Behavioral: Physical activity intervention coupled with standard post-cancer directed treatment care — AYACS will participate in a 16-week physical activity program. AYACS will be instructed to start with a session duration of <15-min, three days per week at low intensity (e.g., activities expending >1.5 to 3 METs or intensity <5 on a scale of 0 to 10). Any type of physical activity will be acceptable. The program will be individualized, and activity increased according to patients' health status, results from the physical function assessment, and most recent week's achieved physical activities. The program will include support calls and texts from research staff (exercise physiologist). The program will be modified and adapted during support calls or texts, including frequency, intensity, time and type to maximize AYACS' success. AYACS will receive a Fitbit at the beginning of the intervention.
  Arms: Physical activity intervention coupled with standard post-cancer directed treatment care group
Other: Standard post-cancer directed treatment care control — AYACS in the control group will not participate in a 16-week physical activity program and will not receive support calls or texts. Physical activity advice according to the Exercise Guidelines for Cancer Survivors will be offered to AYACS following completion of 16-week follow-up. Moreover, AYACS will receive a Fitbit following completion of 16-week follow-up
  Arms: Standard post-cancer directed treatment care control group

SUMMARY:
The purpose of this study is to demonstrate that integration of exercise intervention into standard post-cancer directed treatment care will improve patient reported pain, decrease the need for medications to manage chronic pain and improve functional and psychosocial outcomes in survivors of cancers in adolescents and young adults (AYA). Our central hypothesis is that integration of exercise interventions into standard post-cancer directed treatment care will be acceptable and feasible while improving patients' pain, decreasing the cumulative dose of pain medication and improving patients' functional and psychosocial outcomes as compared to patients who only receive standard post-cancer directed treatment care.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female AYA cancer survivors diagnosed with any type of cancer between the ages of 15 and 39 years old
2. AYA cancer survivors who have completed all standard/planned cancer treatment and are stable at the time of recruitment
3. AYA cancer survivors are < 1-year post cancer therapy
4. AYA cancer survivors who have chronic pain (pain will be self-reported by the participant, will have to be ≥1 on a scale of 10 and lasting for 3 months or longer)
5. AYA cancer survivors who are age ≥18 years old at the time of enrollment
6. AYA cancer survivors who are and who are not non-ambulatory/wheelchair bound.
7. AYA cancer survivors must be able to speak, read and understand the English language
8. AYA cancer survivors must be able to provide and understand informed consent
9. AYA cancer survivors must be able to attend three visits (baseline, 8 and 16-week follow-up) at the Penn State Health Milton S. Hershey Medical Center
10. AYA cancer survivors must have access to a computer with wifi, smartphone with wifi or tablet with wifi

Note: The agreement of the attending oncologist will be required for the participation of AYA cancer survivors eligible for this study.

Exclusion Criteria:

1. AYA cancer survivors who have not completed all standard/planned cancer treatment and/or not in complete remission at the time of recruitment
2. AYA cancer survivors who are > 1-year post cancer therapy
3. AYA cancer survivors who are < 18 years old at the time of enrollment
4. cancer survivors who have evidence of an absolute contraindication to complete any of the physical assessments in their medical record. This exclusion criterion is at the oncologist's discretion when research staff will contact the medical oncologist via secure email or secure message through the electronic medical record for approval to approach their patients for the study and for medical clearance. The oncologists can update this information at any time during the study if there is evidence of an absolute contraindication to complete any of the physical assessments.
5. AYA cancer survivors who have history of refractory or recurrent cancer
6. AYA cancer survivors who are unable to speak, read, and understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | Baseline
  The number of participants approached who agree to participate in the study
Feasibility of the intervention | Baseline to week 16
  The number of participants randomized to the physical activity program intervention coupled with standard post-cancer directed treatment care who complete at least 50% of the physical activity intervention

SECONDARY OUTCOMES:
Measure changes in chronic pain levels | Baseline, week 8 and week 16
  Self-reported chronic pain questionnaire using the Brief Pain Inventory Range 0 to 10, Higher scores indicate more pain and greater interference
Measure changes in cumulative dose of pain medications | Baseline, week 4, week 8, week 12 and week 16
  Chart review: number of pain medications prescribed, total dosage and length of time prescribed.
  Self-reported pain medication: usage of prescription medication and information about the use of non-prescription pain medications (e.g., over the counter oral and topical pain medications).
  The Prescription Drug Monitoring Program will be accessed to gather information on all filled prescriptions for controlled substances within the state of Pennsylvania.
  Morphine equivalent dose will be calculated for each patient after looking at the total daily amount of each opioid the patient is taking. Using the standard conversion factors developed by the CDC, the Morphine milligram equivalent equates the many different opioids into a standard value that is based on morphine and its potency providing an easily interpretable metric for representing opioid utilization
Measure changes in patient reported outcomes | Baseline, week 8 and week 16
  Psychosocial questionnaires using the NIH developed PROMIS questionnaires, including self-reported physical function mobility, anxiety, depressive symptoms, fatigue, social isolation, pain interference, pain intensity, sleep disturbance, sleep-related impairment and cognitive function PROMIS questionnaires assessing patient-reported outcomes on 5-point Likert scale (min value: 1 to max value: 5) responses
Measure changes in physical activity level (Godin-Shephard leisure-time physical activity questionnaire) | Baseline, week 8 and week 16
  Self-reported physical activity questionnaire using the Godin-Shephard leisure-time physical activity questionnaire.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Measure changes in physical activity level (International Physical Activity Questionnaire-Short Form) | Baseline, week 8 and week 16
  Self-reported physical activity questionnaire using the International Physical Activity Questionnaire-Short Form
  * Self-reports physical activity frequency
  * Self-reports physical activity intensity
  * Self-reports physical activity time
  * Self-reports physical activity type
Measure changes in patient functional outcomes (6-min walking test) | Baseline and week 16
  Validated physical function tests, including the 6-min walking test Further distances indicate greater physical function
Measure changes in patient functional outcomes (30-second chair stand test) | Baseline and week 16
  Validated physical function tests, including the 30-second chair stand test Greater amounts of sit/stands indicate greater physical function
Measure changes in patient functional outcomes ("Timed Up and Go" test) | Baseline and week 16
  Validated physical function tests, including the "Timed Up and Go" test Shorter durations indicate greater physical function
Measure changes in patient functional outcomes (grip strength test) | Baseline and week 16
  Validated physical function tests, including the grip strength test Greater grip strength indicate greater physical function

CONTACTS AND LOCATIONS:
Overall Officials: Smita Dandekar, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Health Children's Hospital, Hershey, Pennsylvania, United States